CLINICAL TRIAL: NCT06333210
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Study of the Efficacy and Safety of BCD-180 in Patients With Active Axial Spondyloarthritis
Brief Title: Study of the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of BCD-180 in Patients With Axial Spondyloarthritis (LEVENTA)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-180-3
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Axial Spondyloarthritis
Keywords: biologics; axial spondyloarthritis; monoclonal antibodies; TRBV9
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- bDMARDs and/or tsDMARD experienced subjects, BCD-180 group (Experimental): Subjects in this arm will receive a fixed dose of BCD-180 infusions
  Interventions: Biological: anti-TRBV9 monoclonal antibody infusions
- bDMARDs and/or tsDMARD experienced subjects, Placebo group (Placebo Comparator): Subjects in this arm will receive Placebo infusions till the assessment of the primary endpoint and then will be switched to BCD-180 infusions
  Interventions: Other: Placebo infusions
- bDMARDs and tsDMARD-naive subjects, BCD-180 group (Experimental): Subjects in this arm will receive a fixed dose of BCD-180 infusions and subcutaneous injections of placebo to maintain blindness of adalimumab therapy till the assessment of the primary endpoint, thereafter subjects will receive only BCD-180 infusions
  Interventions: Biological: anti-TRBV9 monoclonal antibody infusions; Other: Placebo subcutaneous injection
- bDMARDs and tsDMARD-naive subjects, Placebo group (Placebo Comparator): Subjects in this arm will receive Placebo infusions and subcutaneous injections of placebo to maintain blindness of adalimumab therapy till the assessment of the primary endpoint, thereafter subjects will be switched to BCD-180 infusions
  Interventions: Other: Placebo infusions; Other: Placebo subcutaneous injection
- bDMARDs and tsDMARD-naive subjects, Adalimumab group (Active Comparator): Subjects in this arm will receive subcutaneous injections of adalimumab and infusions of placebo till the assessment of the primary endpoint, thereafter subjects will be switched to BCD-180 infusions
  Interventions: Other: Placebo infusions; Drug: Adalimumab subcutaneous injection

INTERVENTIONS:
Biological: anti-TRBV9 monoclonal antibody infusions — infusions
  Other Names: BCD-180 infusions
  Arms: bDMARDs and tsDMARD-naive subjects, BCD-180 group; bDMARDs and/or tsDMARD experienced subjects, BCD-180 group
Other: Placebo infusions — infusions
  Arms: bDMARDs and tsDMARD-naive subjects, Adalimumab group; bDMARDs and tsDMARD-naive subjects, Placebo group; bDMARDs and/or tsDMARD experienced subjects, Placebo group
Drug: Adalimumab subcutaneous injection — subcutaneous injection
  Arms: bDMARDs and tsDMARD-naive subjects, Adalimumab group
Other: Placebo subcutaneous injection — subcutaneous injection
  Arms: bDMARDs and tsDMARD-naive subjects, BCD-180 group; bDMARDs and tsDMARD-naive subjects, Placebo group

SUMMARY:
The aim of the study is to evaluate the efficacy, safety, immunogenicity, pharmacokinetics and pharmacodynamics of a fixed dose of study drug (BCD-180) in comparison with placebo in patients with active axial spondyloarthritis (axSpA). The study will include HLA-B27+ patients with radiographic (r-axSpA) and non-radiographic (nr-axSpA) who had no response to prior therapy with non-steroidal anti-rheumatic drugs (NSAIDs), have not received biologic disease-modifying anti-rheumatic drugs (bDMARDs) or targeted synthetic disease-modifying antirheumatic drugs (tsDMARDs), and subjects with insufficient efficacy and/or loss of efficacy on bDMARDs and/or tsDMARDs.

DETAILED DESCRIPTION:
Subjects meeting the eligibility criteria will be randomized in 2 groups:bDMARDs and/or tsDMARD naive subjects and bDMARDs and/or tsDMARD experienced subjects will be randomized independently of each other.

bDMARDs and tsDMARD-naive subjects (naïve) will be randomized into 3 groups:

* BCD-180 (naïve);
* Placebo (naïve);
* Adalimumab.

bDMARDs and/or tsDMARD experienced subjects (exp) will be randomized into 2 groups:

* BCD-180 (exp);
* Placebo (exp).

After the primary endpoint assessment all subjects will be switched to BCD-180.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form for participation in the study.
2. Men and women aged >18 years of age at the time of signing the Informed Consent Form for participation.
3. Positive test result for HLA-B27.
4. 4. Presence of r-axSpA OR nr-axSpA according to the criteria provided below:

   * r-axSpA: axSpA diagnosis meets the ASAS 2009 criteria subject to the presence of radiographic signs of sacroiliitis according to the modified New York criteria (van der Linden et al. 1984) according to the central review. Subjects with an established diagnosis of ankylosing spondylitis according to the modified New York criteria may also be included in the study (van der Linden et al. 1984).
   * nr-axSpA: axSpA diagnosis meets ASAS 2009 criteria in the absence of radiographic signs of sacroiliitis according to the modified New York criteria (van der Linden et al. 1984) according to the central review.
5. Active disease at the screening and the randomization visit diagnosed based on both criteria:

   * ASDAS-CRP ≥2.1
   * assessment of the severity of back pain ≥4 on the NRS (BASDAI, question No. 2).
6. For subjects with nr-axSpA: presence of objective MRI signs of sacroiliitis (according to ASAS/OMERACT) as assessed by the central review AND/OR based on hsCRP level >1.5 ULN at screening.
7. For subjects with r-axSpA: hsCRP level ˃1.5 ULN at screening.
8. Duration of back pain ≥3 months, age <45 years at the onset of the axSpA-associated back pain.
9. Meeting at least one of the following criteria based on the Investigator's assessment:

   * Inadequate response to therapy with NSAIDs defined as insufficient response to therapy with NSAIDs at therapeutic doses for at least 4 weeks, or insufficient response to therapy with two NSAIDs at the maximum permitted dose with the total duration of therapy of at least 4 weeks;
   * Contraindications for therapy with NSAIDs;
   * Intolerance of therapy with more than one NSAID.
10. For bDMARDs-experienced and/or targeted synthetic DMARD-experienced subjects (tsDMARD): meeting at least one of the following criteria based on the Investigator's assessment:

    * lack and/or loss of efficacy, according to the European Alliance of Associations for Rheumatology 2022 (EULAR 2022) recommendations, while on therapy with adequate doses of bDMARDs or tsDMARDs for ≥12 weeks;
    * intolerance of bDMARDs and/or tsDMARDs used for the treatment of axSpA (regardless of treatment duration).
11. For subjects continuing to receive NSAIDs or COX-2 inhibitors: the drug dose shall be steady for at least 14 days prior to Visit 1/Week 0.
12. For women: negative pregnancy test result at screening (the test is not performed in women who have been postmenopausal for at least 2 years or are surgically sterile) .
13. The ability of the subject to follow the Protocol procedures, according to the Investigator.
14. Willingness of subjects and their sexual partners of childbearing potential to use reliable methods of contraception from the date of signing the ICF, throughout the study, and for 8 weeks after the last administration of BCD-180/placebo (infusions)/adalimumab/placebo (subcutaneously). This requirement does not apply to subjects who have had operative sterilization and women who have been postmenopausal for more than 2 years.
15. For participants of childbearing potential, from signing the informed consent form, throughout the study, and for 8 weeks after the last dose of BCD-180/placebo (intravenously)/adalimumab/placebo (subcutaneous):

    * no egg donation for female subjects;
    * no sperm donation for male subjects.

Exclusion Criteria:

1. Refusal to take NSAIDs for the treatment of axSpA for any subjective reasons that do not have a clinical justification.
2. Use of the following medicines/procedures:

   * at any time before signing the ICF: total lymphoid irradiation;
   * at any time before signing the ICF: bone marrow transplantation, including stem and hematopoietic cell transplantation for any indications;
   * at any time before signing the ICF: splenectomy;
   * within 8 weeks before signing the ICF: treatment with immunoglobulins;
   * within 12 months before signing the ICF: use of immunosuppressants. Exception: glucocorticoids. A subject receiving glucocorticoids may be included in the study provided that the daily dose of glucocorticoids is ≤10 mg/day (calculated with reference to prednisolone) and was stable for at least 4 weeks prior to the Randomization Visit.
   * within 4 weeks before signing the ICF and during the screening period: use of synthetic DMARDs and thiopurines, including, but not limited to: 6-mercaptopurine, azathioprine, and others.

   Exception: the medicinal products listed below if their dose was stable for 4 weeks before signing the ICF and during the screening period:
   * oral or parenteral methotrexate at a dose ≤25 mg/week, therapy shall be started at least 8 weeks before signing the ICF;
   * 5-aminosalicylic acid and its derivatives, including sulfasalazine, at a dose not exceeding 3 g/day, provided that therapy was started at least 8 weeks before signing the ICF. Subjects with inflammatory bowel disease (IBD) may be treated with topical 5-aminosalicylic acid at therapeutic doses;

     * intra-articular and paraspinal glucocorticoids within 4 weeks prior to the Randomization Visit, intramuscular glucocorticoids within 2 weeks prior to the Randomization Visit;
     * use of alkylating agents at any time within 12 months prior to signing the ICF;
     * BCD-180 administration at any time before signing the ICF.
3. Vaccination with any vaccines within 12 weeks prior to signing the ICF.
4. Documented presence of one or more of the listed conditions:

   * within 8 weeks before signing the ICF and during the screening period: exacerbated IBD (attack of Crohn's disease or exacerbation (relapse, attack) of ulcerative colitis), severe, generalized, pustular, exudative, psoriasis of the hands and feet;
   * acute uveitis within less than 2 weeks prior to signing the ICF and during the screening period.

   Clarification: for subjects with IBD: IBD therapy must be stable for 8 weeks prior to signing the ICF. For subjects with psoriasis: topical products may be used.
5. A current diagnosis or a history of a severe immunodeficiency of any origin.
6. A diagnosis of HIV infection, hepatitis B, hepatitis C.
7. The following laboratory test results at screening:

   * Transaminase (ALT and/or AST) activity >1.5×ULN;
   * ALP activity >1.5×ULN;
   * WBC count <3.0 cells×109/L;
   * Neutrophil count <1.5 cells×109/L;
   * Lymphocyte count <0.8 cells×109/L;
   * Platelet count <100 cells × 109/L;
   * Hemoglobin level <100 g/L;
   * Serum blood creatinine >ULN.
8. Clinically significant thyroid disease and/or clinically significant deviation of the TSH level from the reference values at screening.
9. Diagnosis of active or latent tuberculosis, including a history of tuberculosis .
10. Major surgery within 4 weeks prior to signing the ICF or major surgery planned for the period of participation in the study.
11. Documented diagnosis of infectious mononucleosis within 8 weeks prior to signing the ICF and during the screening period, any active infection or recurrent infection within 4 weeks prior to signing the ICF and during the screening period, including fever ≥38°C at the Randomization Visit.
12. Documented diagnosis of any other chronic infection that, in the opinion of the investigator, can increase the risk of infectious complications.
13. Severe infectious diseases (requiring hospitalization, parenteral use of antibacterial, antimycotic or antiprotozoal drugs) within 8 weeks prior to signing the ICF and during the screening period.
14. Systemic antibacterial, antimycotic or antiprotozoal therapy within 8 weeks prior to signing the ICF and during the screening period.
15. Epileptic seizures, a history of seizures.
16. A history of or current (at the time of signing the ICF and during the screening period) significant uncontrolled neuropsychiatric disorders, severe depression and/or suicide attempts, a risk of suicide and/or any psychiatric illness that, in the opinion of the investigator, may pose an excessive risk to the subject or have an impact on the subject's ability to follow the protocol.
17. Known (including from historical data) alcohol or drug dependence, psychoactive substance or drug abuse, evidence of alcohol/drug dependence or current abuse that, in the investigator's opinion, is a contraindication to AS therapy or limits treatment adherence.
18. The following diseases:

    * at screening and/or in the past and at the Randomization Visit: non-axSpA inflammatory joint disease (including rheumatoid arthritis, gout, psoriatic arthritis, Lyme disease, etc.),
    * at screening and/or at the Randomization Visit: reactive arthritis,
    * at screening and/or in the past and at the Randomization Visit: systemic autoimmune diseases (including systemic lupus erythematosus, systemic scleroderma, inflammatory myopathy, mixed forms of inflammatory connective tissue diseases, overlap syndrome, etc.).

    Exception: the following subjects may be included in the study:
    * eligible patients with psoriasis;
    * diagnosed with IBD, at the stage of remission without the need for systemic therapy;
    * with uveitis associated with axSpA, except for subjects with severe visual impairment or with sight in one eye, subjects with corneal opacity, significant cataract, posterior capsule opacity, or posterior synechia in the studied eye of such severity that makes assessment of uveitis severity insufficient or impossible. Clarification: the study may include subjects with prior acute uveitis 2 weeks after the resolution, including those receiving topical therapy, including intra-bulbar administration of glucocorticoids.
19. Comorbidities (including, but not limited to, metabolic, hematological, renal, hepatic, pulmonary, neurological, endocrine, cardiac, infectious, gastrointestinal disorders), including disorders ongoing at the time of screening, which, in the opinion of the investigator, may affect the course of radiographic axSpA, the results of assessment of its symptoms, or create an unacceptable risk to the subject from study therapy.
20. Known allergy or intolerance to any component of the test drug, premedication drugs used in this clinical study. For bDMARDs and/or tsDMARD-naive subjects: known allergy or intolerance of any components of adalimumab.
21. For bDMARDs and/or tsDMARD-naive subjects: contraindications for the use of adalimumab.
22. A history of angioedema.
23. Fibromyalgia, or other conditions associated with chronic pain .
24. Lymphoproliferative diseases or malignancies with a remission duration of less than 5 years, with the exception of cured basal cell carcinoma and cervical cancer in situ.
25. Pregnancy, pregnancy planning (including pregnancy of female sexual partners of male study subjects) less than 8 weeks after the last administration of BCD-180/placebo (intravenously)/adalimumab/placebo (subcutaneous), breastfeeding.
26. Contraindications to MRI.
27. Simultaneous participation in other clinical studies, as well as previous participation in other clinical studies less than 3 months before signing the ICF, prior participation in this study.

Exception: subjects who dropped out of this study at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieved ASAS40 among bDMARDs and tsDMARD-naive subjects | [Time Frame: week 24]
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 40% or more
Proportion of subjects who achieved ASAS40 among bDMARDs and/or tsDMARD-experienced subjects | [Time Frame: week 24]
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 40% or more

SECONDARY OUTCOMES:
Proportion of subjects who achieved ASAS40 among subjects with r-axSpA | [Time Frame: week 24]
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 40% or more
Proportion of subjects who achieved ASAS40 among subjects with nr-axSpA | [Time Frame: week 24]
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 40% or more
Proportion of subjects with the ASDAS-CRP <1.3 | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Proportion of subjects with the Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) score <1.3
Proportion of subjects with the ASDAS-CRP ≥1.3 - <2.1 | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Proportion of subjects with the Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) score ≥1.3 - <2.1
Proportion of subjects with the ASDAS-CRP ≥2.1 - ≤3.5 | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Proportion of subjects with the Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) score ≥2.1 - ≤3.5
Proportion of subjects with the ASDAS-CRP >3.5 | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Proportion of subjects with the Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) score >3.5
Proportion of subjects who achieved ASDAS-CII (clinically important improvement) | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Clinically important improvement defined as a decrease from baseline in ASDAS ≥1.1
Proportion of subjects who achieved ASDAS-MI (Major improvement) | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Major improvement (MI) defined as a decrease from baseline in ASDAS ≥2.0
ASDAS-CRP change from baseline | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
Proportion of patients who achieved clinical response defined as an improvement of BASDAI by at least 50% compared to baseline | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
Change from baseline in BASDAI | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Proportion of subjects who achieved ASAS40 | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 40% or more
Proportion of subjects who achieved ASAS20 | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 20% or more
Proportion of subjects who achieved ASAS5/6 | [Time Frame: weeks 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Ratio of patients who developed a response in at least 5 of 6 criteria of ankylosing spondylitis assessment score (ASAS)
Proportion of subjects who achieved ASAS partial remission | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
Change from baseline in BASMI | [Time Frame: weeks 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Change from baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) score
Change from baseline in BASFI | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) score
Change from baseline in the swollen joint count (44 joints) | [Time Frame: weeks 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
Change from baseline in MASES | [Time Frame: weeks 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Change from baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES)
Change from baseline in overall back pain severity (BASDAI No. 2) | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
Change from baseline in nocturnal back pain severity | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
  Change from baseline in nocturnal back pain score during measured by Visual Analog Scale for Pain
Change in the patient global assessment of disease activity from baseline | [Time Frame: weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156]
Change in the quality of life score assessed with EQ-5D-3L questionnaire from baseline | [Time Frame: weeks 12, 24, 48, 72, 84, 96, 108, 132, 156, 160]
Change from baseline in SF-36 Physical Functioning compared to baseline | [Time Frame: weeks 4, 8, 12, 16, 20, 24, 48, 72, 84, 96, 108, 120, 132, 144, 156, 160]
Change from baseline in SF-36 Mental Health compared to baseline | [Time Frame: weeks 4, 8, 12, 16, 20, 24, 48, 72, 84, 96, 108, 120, 132, 144, 156, 160]
Change in the WPAI score from baseline | [Time Frame: weeks 12, 24, 48, 72, 84, 96, 120, 132, 144, 156, 160]
  Change from baseline in Work Productivity and Activity Impairment (WPAI)
Change in the ASAS HI score from baseline | [Time Frame: weeks 12, 24, 48, 72, 84, 96, 120, 132, 144, 156, 160]
  Change from baseline in ASAS Health Index
Change in the concentration of hsCRP from baseline | [Time Frame: weeks 4, 8, 12, 16, 20, 24, 48, 72, 84, 96, 108, 120, 132, 144, 156, 160]
Change in ESR from baseline | [Time Frame: weeks 4, 8, 12, 16, 20, 24, 48, 72, 84, 96, 108, 120, 132, 144, 156, 160]
Changes in the SPARCC score (spine, SIJ) from baseline | [Time Frame: weeks 24, 48, 108, 144, 156]
  Change from baseline in Spondyloarthritis Research Consortium of Canada Enthesitis (SPARCC)
Changes in mSASSS scores from baseline | [Time Frame: weeks 48, 108, 144,156]
  Change from baseline in Modified stoke ankylosing spondylitis spinal score (mSASSS)
Proportion of subjects with adverse events | [Time Frame: weeks 24, 160]
Proportion of subjects with serious adverse events | [Time Frame: weeks 24, 160]
Proportion of subjects with grade 3 or higher adverse events according to CTCAE 5.0 | [Time Frame: weeks 24, 160]
Proportion of subjects prematurely withdrawn from the study due to adverse events | [Time Frame: weeks 24, 160]

CONTACTS AND LOCATIONS:
Overall Officials: Arina Zinkina-Orikhan, PhD, MD, Study Director — Director of Clinical Development Department, BIOCAD
Locations (32):
- Belarus (2):
  - 1St City Clinical Hospital, Minsk, Minsk
  - State Institution "Minsk Scientific and Practical Center for Surgery, Transplantology and Hematology", Minsk
- Russia (30):
  - KGBU "City Hospital No. 4 named after N.P. Gull, Barnaul", Barnaul
  - Chelyabinsk Regional Clinical hospital, Chelyabinsk
  - Regional State Budgetary Healthcare Institution "Irkutsk City Clinical Hospital 1", Irkutsk
  - Republican Clinical Diagnostic Center of the Ministry of Health of the Udmurt Republic, Izhevsk
  - Republican Clinical Hospital of the Ministry of Health of the Republic of Tatarstan, Kazan'
  - State Autonomous Healthcare Institution "Kuzbass Clinical Emergency Hospital named after M. A. Podgorbunsky", Kemerovo
  - Federal State Budgetary Institution "Pirogov National Medical Surgical Center" of the Ministry of Health of the Russian Federation, Moscow
  - Federal State Budgetary Scientific Institution "Research Institute of Rheumatology named after V.A. Nasonova", Moscow
  - State Budgetary Healthcare Institution of Moscow City "City Clinical Hospital 15 named after O.M. Filatov of the Moscow City Health Department", Moscow
  - State Budgetary Healthcare Institution of Moscow City Clinical Hospital 1 named after N.I. Pirogov of the Moscow City Health Department, Moscow
  - State Budgetary Higher Vocational Education Institution I.M. Sechenov First Moscow State Medical University, Moscow
  - State Budgetary Healthcare Institution "Center of Allergology and Immunology" of Kabardino-Balkarian Republic, Nal'chik
  - State Budgetary Healthcare Institution of the Nizhny Novgorod Region "Nizhny Novgorod Regional Clinical Hospital named after N. A. Semashko", Nizhny Novgorod
  - Federal State Budgetary Scientific Institution "Institute of Cytology and Genetics of the Siberian Branch of the Russian Academy of Sciences", Novosibirsk
  - Budgetary healthcare institution of the Omsk region "Regional clinical hospital", Omsk
  - State Budgetary Healthcare Institution of Perm Krai "Order of Honour" Perm Regional Clinical Hospital ", Perm
  - Federal State Budgetary Educational Institution of Higher Education "Rostov State Medical University" of the Ministry of Health of the Russian Federation, Rostov-on-Don
  - Clinical Rheumatology Hospital №25, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "St. Petersburg State University", Saint Petersburg
  - Federal State Budgetary Institution "Almazov National Medical Research Center" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - North-Western State Medical University n.a. I.I.Mechnikov, Saint Petersburg
  - State Budgetary Healthcare Institution "Samara Regional Clinical Hospital named after V.D. Seredavin", Samara
  - Private Healthcare Institution "Clinical Hospital" RD-Medicine "of the city of Saratov, Saratov
  - Private Healthcare Institution "Clinical Hospital" RD-Medicine "of Smolensk, Smolensk
  - Federal State Budgetary Educational Institution of Higher Education "Siberian State Medical University", Tomsk
  - Republican Clinical Hospital named after G. G. Kuvatov, Ufa
  - State Healthcare Institution Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - State Healthcare Institution "City Clinical Emergency Hospital 25", Volgograd
  - State Budgetary Healthcare Institution of the Yaroslavl Region "Clinical Hospital named after N.A. Semashko", Yaroslavl
  - State Autonomous Healthcare Institution of the Sverdlovsk Region "City Clinical Hospital 14 Ekaterinburg", Yekaterinburg